CLINICAL TRIAL: NCT06229080
Title: Short-term Embolization Using Gelatin Particles for FloW ModulAtion During Y90 Radioembolization
Acronym: SEGWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GuardGel NXG001
Record Dates: First submitted 2024-01-05; First posted 2024-01-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Liver Cancer (Primary and Metastatic)
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): short-acting gelatin sponge particles (NexGel) will be administered to the hepatic arteries toward the non-tumorous liver.
  Interventions: Device: NexGel

INTERVENTIONS:
Device: NexGel — When a planned perfused area includes two or more Couinaud segments and more than 50% of the target area is non-tumorous liver, short-acting gelatin sponge particles (NexGel) will be administered to the hepatic arteries toward the non-tumorous liver. The embolization particles will be prepared by mixing one vial of the particles with 5 mL of iodinated contrast agents and intra-arterially delivered with a microcatheter 2.0-Fr or larger. After confirming the disappearance or substantial reduction of liver parenchymal staining of the embolized area on angiography, radioembolization using Y90 glass or resin microspheres will be conducted. Digital subtraction angiography will be performed 30 minutes after the transient embolization to identify recanalization of the transiently embolized hepatic arteries.

SUMMARY:
The SEGWAY trial is a prospective, single-arm clinical study to evaluate the efficacy and safety of flow diversion to protect non-tumorous liver function using short-acting gelatin sponge particles during Yttrium-90 radioembolization of liver cancer.

DETAILED DESCRIPTION:
Short-acting gelatin sponge particles will be used during radioembolization to protect normal liver tissue in patients with liver cancer whose treatment field encompasses a substantial portion of non-tumorous liver tissue. Recanalization of the embolized hepatic artery will be assessed by angiography within 30 minutes following the procedure. Suppression of Y90 microsphere delivery to the protected, non-tumorous liver tissue will be evaluated using Y90 PET-CT imaging, by comparing the protected regions to non-protected, non-tumorous regions within the perfused area. Enhanced tumor uptake of Y90 microspheres will be quantified using the tumor-to-normal liver ratio (TNR), calculated by comparing pre-procedure SPECT-CT with post-procedure PET-CT data. Finally, preservation of liver function in protected tissue relative to unprotected tissue will be assessed six months post-procedure using signal intensity ratios on hepatobiliary phase images obtained from gadoxetic acid-enhanced MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older
2. Patients diagnosed with primary or metastatic liver cancer based on histological and/or radiological findings
3. Patients determined, following medical, surgical, or multidisciplinary evaluation, to be best treated by radioembolization
4. Patients with no history of local treatments (e.g., ablation, chemoembolization) to the same hepatic lobe within the past year
5. Child-Pugh class A
6. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or lower
7. Patients whose treatment area, as determined by planning angiography, includes at least two liver segments
8. Patients for whom normal liver tissue constitutes 50% or more of the treatment volume

Exclusion Criteria:

1. Liver cancer with vascular invasion
2. For primary liver cancer, patients who have been diagnosed with a malignancy other than the primary liver cancer within 2 years prior to study enrollment
3. Patients who have undergone biliary-enteric anastomosis
4. Patients with an estimated lung dose of 30 Gy or higher on pre-procedure 99mTc-MAA imaging
5. Patients with a known contraindication to gelatin use

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Mean absorbed dose ratio between the protected perfused liver and unprotected perfused liver | Day 1, The day after radioembolization
  Mean absorbed dose ratio between the protected perfused liver and unprotected perfused liver

SECONDARY OUTCOMES:
Angiographic recanalization of the transiently embolized hepatic arteries | After Y-90 microsphere infusion, 30 minutes after embolization
  Angiographic recanalization of the transiently embolized hepatic arteries (grade 0, completely occluded; grade 1, antegrade flow visible only near the RGM injection point; grade 2, sluggish antegrade flow visible to the periphery; and grade 3, completely patent)
Tumor-to-normal liver ratio change between the pre-treatment SPECT-CT (99mTc-MAA injection without transient embolization) and post-treatment PET-CT (Y90 injection with transient embolization) | Day 1, The day after radioembolization
  Tumor-to-normal liver ratio change between the pre-treatment SPECT-CT (99mTc-MAA injection without transient embolization) and post-treatment PET-CT (Y90 injection with transient embolization)
Ratio of the Relative volumetric changes between the protected perfused liver and unprotected perfused liver | 6 months after radioembolization
  Ratio of the Relative volumetric changes between the protected perfused liver and unprotected perfused liver
Relative signal intensity ratio between the protected perfused liver and unprotected perfused liver on a 20-minute delayed scan of gadoxetic acid-enhanced MRI | 6 months after radioembolization
  Relative signal intensity ratio between the protected perfused liver and unprotected perfused liver on a 20-minute delayed scan of gadoxetic acid-enhanced MRI
Response to the treatment, as assessed by mRECIST | 6 months after radioembolization
  Objective Tumour Response will be assessed by the investigators on CT/MRI image analysis
Serious adverse event | For 6 months from radioembolization
  Serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Choi, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea